CLINICAL TRIAL: NCT00686127
Title: A Randomized, Double-Blind, Placebo-Controlled Trial (RDBPCT) of the Effectiveness of the Lidocaine Patch in the Management of Neuropathic Pain After Breast Cancer Surgery
Brief Title: Symptom Management After Breast Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Breast Pain; CA107091
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2014-04

CONDITIONS: Neuropathic Pain; Postmastectomy Pain
Keywords: breast cancer; neuropathic pain; topical lidocaine; postmastectomy pain; breast symptoms; breast pain
MeSH Terms: conditions — Neuralgia; Breast Neoplasms; Mastodynia | interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine Patch (Active Comparator): Drug: lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.), 1 patch was applied topically to the affected site(s) for 12 hours each day.
  Interventions: Drug: Lidoderm patch
- Placebo Patch (Placebo Comparator): Drug: placebo patch, 1 patch was applied topically to the affected site(s) for 12 hours each day.
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Lidoderm patch — 1 patch was applied topically to the affected site(s) for 12 hours each day.
  Other Names: Lidoderm, Lidoaine patch 5%
  Arms: Lidocaine Patch
Drug: Placebo patch — 1 patch was applied topically to the affected site(s) for 12 hours each day.
  Arms: Placebo Patch

SUMMARY:
This trial is part of a larger, longitudinal study of symptoms that occur in the breast surgical scar area and/or ipsilateral arm following breast cancer surgery. Women who develop pain in the breast scar area or ipsilateral arm will be randomized to a placebo patch or a lidocaine patch that they will wear on a daily basis for 12 weeks. We hypothesize that women who wear the lidocaine patch will report a decrease in pain and decreased interference with function compared to women who wear the placebo patch.

ELIGIBILITY:
Inclusion Criteria:

* Adult women >18 years who develop neuropathic pain in the breast scar area and/or ipsilateral arm following breast cancer surgery
* Has a healed incision(s)
* Has no recurrent disease in the painful area
* Is able to read, write and understand English

Exclusion Criteria:

* Presence of another type of pain that is more severe than the neuropathic pain
* Use of an opioid analgesic of greater than 60 mg codeine/day
* Is actively trying to become pregnant
* Has a medical contraindication to the use of lidocaine
* Has an allergy to lidocaine
* Is taking a coanalgesic for neuropathic pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Patch: Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.), 1 patch was applied topically to the affected site(s) for 12 hours each day.
Period: Overall Study
Arm/Group | Lidocaine Patch | Placebo Patch
Started | 14 | 7
Completed | 0 (Patients withdrew from the study because they did not like wearing the patch.) | 1
Not Completed | 14 | 6
Not completed — Withdrawal by Subject | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine Patch: Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.): 1 patch was applied topically to the affected site(s) for 12 hours each day.
- Total: Total of all reporting groups
Arm/Group | Lidocaine Patch | Placebo Patch | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.3) | 46.1 (13.5) | 49.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9 | 2 | 11
  Black | 3 | 0 | 3
  Asian/Pacific Islander | 1 | 3 | 4
  Hispanic or Mixed Ethnic Background | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 7 | 21
Average pain intensity [Mean (Standard Deviation); unit: units on a scale] — Patients scored their pain intensity in the breast and/or ipsilateral arm at enrollment using a 0 to 10 numeric rating scale, ranging from no pain (0) to worst pain imaginable (10)
  units on a scale | 5.3 (2.3) | 4.2 (1.1) | 4.8 (1.9)
Worst pain intensity [Mean (Standard Deviation); unit: units on a scale] — Patients scored their pain intensity in the breast and/or ipsilateral arm at enrollment using a 0 to 10 numeric rating scale, ranging from no pain (0) to worst pain imaginable (10)
  units on a scale | 7.8 (1.5) | 6.4 (4.8) | 7.1 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity on an 11-point Scale From Baseline to 12 Weeks
Description: Patients scored their pain intensity in the breast and/or ipsilateral arm using a 0 to 10 numeric rating scale, ranging from no pain (0) to worst pain imaginable (10). The change in pain intensity was calculated from two time points as the later time point (12 weeks) minus the earlier time point (Baseline).
Time Frame: Baseline, 12 weeks
Population: This study attempted to evaluate changes in average pain intensity following breast cancer surgery. However, since none of the patients in the lidocaine group completed the 12 week trial, the outcomes of this study cannot be evaluated.
Measure: Number; unit: units on a scale
Arm/Group | Lidocaine Patch | Placebo Patch
Number analyzed (Participants) | 0 | 1
units on a scale |  | 4.0 (0.0)

2. Secondary Outcome: Pain Interference With Function
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Lidocaine Patch: Lidocaine patch One patch is changed every twenty-four hours
- Placebo Patch: Placebo patch: Patch is changed every 24 hours
Arm/Group | Lidocaine Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 0/14 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes